CLINICAL TRIAL: NCT00963391
Title: "Alcohol Based Hand Sanitizers for the Prevention of Acute Diarrheal Disease and Acute Respiratory Infection in Children Under 5 Attending Childcare Centers in Bogotá, Cundinamarca and Tolima, in Colombia: a Cluster Randomized Control Trial"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Collaborators: Fedesarrollo (Unknown); Pontificia Universidad Javeriana (Other); Global Development Network (Unknown)
Responsible Party: Juan C. Correa/Director of the Community Health Division, Fundación Santa Fe de Bogotá
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TMPCOL298
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Acute Diarrheal Disease; Acute Respiratory Infection
Keywords: Health Production; Government Policy; Regulation; Public Health; Government Policy; Provision and Effects of Welfare Programs; Gastrointestinal diseases; Respiratory Tract Infections; Diarrhea; Ethanol; Child, Preschool; Handwashing
MeSH Terms: conditions — Gastrointestinal Diseases; Respiratory Tract Infections; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABHS use (Experimental): Centers assigned to the intervention group were provided with ABHS dispensers with a gel solution with ethyl alcohol at 62% as active ingredient (Purell®, GOJO Industries, Dayton, Ohio). Proper safety measures were followed. Standardized ABHS training workshops for staff and children in centers allocated to the intervention were carried out simultaneously with dispenser installation. Thirty minute refresher sessions about ABHS technique were provided to staff and children on a monthly basis, for a total of 8 sessions per center.
  Interventions: Other: ABHS use
- No treatment (No Intervention): Centers assigned to the control group received no hand hygiene recommendations other than to continue with current hand hygiene practices and no further information on hand hygiene other than the general information received before trial initiation was provided.

INTERVENTIONS:
Other: ABHS use — Centers assigned to the intervention group were provided with ABHS dispensers with a gel solution with ethyl alcohol at 62% as active ingredient (Purell®, GOJO Industries, Dayton, Ohio). A total of 85 dispensers were installed, one dispenser was installed in each center of size less than 14 children, and one per classroom plus an additional one for common areas in centers with more than 28 children. Proper safety measures were followed.
  Standardized ABHS training workshops for staff and children in centers allocated to the intervention were carried out simultaneously with dispenser installation. Thirty minute refresher sessions about ABHS technique were provided to staff and children on a monthly basis, for a total of 8 sessions per center.
  Other Names: Purell®, GOJO Industries, Dayton, Ohio
  Arms: ABHS use

SUMMARY:
The purpose of this study is to conduct a Randomized Control Trial (RCT) in a developing country setting in order to evaluate the role of alcohol based hand sanitizers (ABHS) in preventing the transmission of infectious diseases in areas where water is a scarce resource. The investigators want to find out if the use of ABHS reduces the incidence of two leading causes of morbidity and mortality in children under 5 years of age in the developing world: acute diarrheal disease (ADD) and acute respiratory infections (ARI).

DETAILED DESCRIPTION:
We performed a cluster, RCT in child care centers located in six urban settings of Colombia with intermittent tap water availability. A total of 1727 children between 1 and 5 years of age distributed in 42 childcare centers participated in the study. The intervention consisted on installation of ABHS gel dispensers and training on their use by participating children in child care centers. Centers assigned to the control group were recommended to continue with current hand hygiene practices. Child care centers matched by location, size and sanitary conditions were randomly assigned to intervention or control. Cases of Acute Diarrheal Disease (ADD) and Acute Respiratory Infections ARI were identified through teacher reported signs and symptoms of disease and validated by a trained physician. We also monitored adverse events potentially related to ABHS. To compare incidence rates between study arms we modeled the number of episodes of ADD and ARI per child using a Cox proportional hazards multiple regression with random effects.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 and 5 years of age
* Attending child care centers with limited tap water availability

Exclusion Criteria:

* Chronic conditions
* Not willing to participate

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1727 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Number of Cases of Acute Diarrheal Disease Number of Cases of Acute Respiratory Infection | April - December 2008

SECONDARY OUTCOMES:
Number of Adverse Events | April - December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Correa, MD, Principal Investigator — Fundación Santa Fe de Bogotá; Diana Pinto, MD, Principal Investigator — Fedesarrollo, Pontificia Universidad Javeriana
Locations (1):
- Fundación Santa Fe de Bogotá, Bogotá, D.C., Colombia